CLINICAL TRIAL: NCT06430281
Title: Development and Pre-testing of a Manual Therapy Force Perception Scale
Brief Title: Manual Therapy Force Perception Scale
Status: Completed | Type: Observational
Sponsor: Université du Québec à Trois-Rivières (Other)
Responsible Party: Principal Investigator, Isabelle Pagé, Professor, Université du Québec à Trois-Rivières
Other Study IDs: UQTR_IP_EchelleTM_2024
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Manual Therapy
Keywords: Chiropractic; Spinal mobilization; Spinal manipulation; force sensor
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants: Chiropractors will administer manual therapies on a manikin utilizing three distinct levels of force (typical force, low force, high force), determined by the trial label on the scale. A sensor will gauge the magnitude of force applied.
  Interventions: Other: Manual therapy

INTERVENTIONS:
Other: Manual therapy — A manual force will be applied to a manikin positioned on a chiropractic treatment table. The force exerted during the manual therapy must align with the trial label indicated on the Manual Therapy Force Perception [MTFP] scale.

SUMMARY:
The objective of this observational study is to pilot a scale designed to assist clinicians in evaluating the force they perceive during manual therapy.

The main question it aims to answer is:

- Are clinicians able to evaluate the force they use when delivering manual therapies to their patients using a scale?

For the pilot test, licensed chiropractors administer manual therapies on a manikin.

DETAILED DESCRIPTION:
The aim of this observational study is to pilot test an ordinal scale (the Manual Therapy Force Perception [MTFP] scale) intended to enable clinicians to assign ordinal rankings to their patients based on their perception of the force they applied during manual therapy . This involved evaluating the agreement between the force applied by clinicians during spinal manipulations and mobilizations delivered on a manikin and their subjective perception of force, as determined using the MTFP scale. Additionally, the pilot study aimed to seek feedback on the MTFP scale from clinicians who are its potential users.

ELIGIBILITY:
Inclusion Criteria:

* Licensed chiropractors with a private practice within the province of Quebec, Canada.

Exclusion Criteria:

* Having a condition that prevents the execution of approximately 50 manual therapies over a 1-hour period.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Licensed chiropractors
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Peak force measured by a force sensor during the manual therapy | During the manual therapy
  The therapy will be delivered on a force sensor (Loadpad(R)) which will measured the force applied. The peak force reached during the therapy will be extracted.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Pagé, DC, PhD, Principal Investigator — Université du Québec à Trois-Rivières
Locations (1):
- Université du Québec à Trois-Rivières, Trois-Rivières, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No